CLINICAL TRIAL: NCT01931579
Title: Assessment of Probe Based Confocal Laser Endo-microscopy for In-vivo Diagnosis of Peripheral Lung Nodules and Masses. "NODIVEM" Study
Brief Title: Assessment of Probe Based Confocal Laser Endo-microscopy for In-vivo Diagnosis of Peripheral Lung Nodules and Masses.
Acronym: NODIVEM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011/103/HP; 2011-AO1053-38 (Other: RCB)
Record Dates: First submitted 2013-07-29; First posted 2013-08-29 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Nodule Persistent; Malignant Neoplasm of the Respiratory System; Benign Neoplasms of the Respiratory System
Keywords: confocal endo-microscopy, lung nodule, respiratory neoplasms
MeSH Terms: conditions — Respiratory Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- confocal endo-microscopy (Experimental): confocal endo-microscopy : CELLVIZIO endo-microscopy procedure is performed in every patient using the same extended working channel as for navigational bronchoscopy.
  Interventions: Device: confocal endo-microscopy

INTERVENTIONS:
Device: confocal endo-microscopy — The intervention consists of the use of confocal endo-microscopy using the CELLVIZIO device and either the 1 mm CELLVIZIO miniprobe (ALVEOFLEX) or the 0.6 mm CELLVIZIO miniprobe (CHOLANGIOFLEX), during a navigational bronchoscopy procedure for the diagnostic of peripheral nodule. In this study, the navigational device - either radial endobronchial ultrasound (EBUS) or electromagnetic navigation (EMN) - will be moved to another location if the CELLVIZIO displays a non solid pattern, indicating that the nodule may not have been reached during the procedure. Three attempts of EBUS or EMN are allowed until the CELLVIZIO shows a solid pattern.
  Other Names: CELLVIZIO Lung 488 nm and 660 nm; 1 mm CELLVIZIO miniprobe (ALVEOFLEX); 0.6 mm CELLVIZIO miniprobe (CHOLANGIOFLEX)

SUMMARY:
Solitary pulmonary nodule has become a major challenge in respiratory clinical practice. According to published guidelines, their management often requires close CT follow up, PET CT and invasive procedures to obtain a definite histology. In this context, innovative endoscopic techniques refered as navigational bronchoscopy have proved to be efficient, for the localization and sampling of peripheral lung nodules. However, these techniques are unable to differentiate malignant lesions from benign ones, in-vivo, in real time. Confocal endo-microscopy (CELLVIZIO) of the distal lung - also refered as distal lung probe based confocal laser endo-microscopy or alveolar lung endo-microscopy - allows in-vivo imaging of the distal lung structures in real time.

This prospective trial we will assess confocal endoscopy as a tool to localize the peripheral lung nodules and to differentiate benign from tumoral lesions.

Objective(s)

1. To demonstrate that confocal endo-microscopy is not inferior to navigational endoscopy for the localisation of peripheral lung nodule
2. To demonstrate that confocal endoscopy can differentiate benign from malignant tumors

Experimental design:

Multicentric prospective controlled trial, conducted in three academic centers, specialized in interventional bronchoscopy, equipped with both navigational bronchoscopy and probe based confocal endo-microscopy.

Subjects with peripheral lung nodule requiring navigational bronchoscopy will be explored using both Confocal endoscopy AND navigational bronchoscopy. Confocal probe will be inserted in the same catheter as used for the navigational bronchoscopy and confocal images will be recorded before sampling. An ancillary study using topical methylene blue as in situ will be conducted at the Rouen University Center.

An ancillary protocol includes the use of in situ methylene blue deposition and 660 confocal endo-microscopy analysis.

DETAILED DESCRIPTION:
Main assessment criteria:

1. number of lesions localized by confocal endoscopy compared to navigational bronchoscopy
2. Positive and negative predictive values of confocal signs before and after IV fluorophore injection for the diagnosis of cancer.

In this this study, positive diagnostic criteria for the localization of peripheral nodule using confocal imaging is a solid pattern as opposed to the usual loose fibered network pattern of the normal alveolar duct. According to this criteria, the confocal imaging procedure will be considered as valid if the number of lesions localized by confocal is not inferior to 90 % of those localized by navigational bronchoscopy. Therefore, probe based confocal laser endo-microscopy will prove valid if it can recognize at least 70 subjects out of the 78 / 120 subjects for which the navigational bronchoscopy is forecasted to localize the peripheral lesion (Cohen concordance Kappa value of 0,74 between confocal and navigational bronchoscopy).

A secondary objective will be to describe specific signs of cancer using confocal endoscopy . This will be assessed on the first 30 patients using confocal imaging obtained before and after fluorophore IV injection, in comparison to histology, and confirmed on the following 48 patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a peripheral lung nodule accessible by navigational bronchoscopy and CELLVIZIO according to Investigator evaluation of the CT scan.
* 18 years old or more.
* Affiliation to french social security insurance.
* Signed informed consent for the procedure.

Exclusion Criteria:

* Severe respiratory insufficiency that will not allow the bronchoscopy procedure
* Uncorrected bleeding disorders
* History of pneumonectomy or exploration controlateral to a non functional lung,
* Pregnant or breast feeding woman, or person not authorized to participate to a clinical trial according to L1121-6 et L1121-8 of French Code of Public Health, concurrent participation to another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-05; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity of confocal imaging (solid pattern) for the diagnostic of the pulmonary nodule | six months after the procedure
  Confocal imaging will be considered as "positive" when both
  * a solid pattern is displayed
  * a diagnostic biopsy is obtained at the site of confocal imaging

CONTACTS AND LOCATIONS:
Overall Officials: Luc C Thiberville, MD, Principal Investigator — University Hospital, Rouen
Locations (3):
- France (3):
  - UHRouen, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - CHU Toulouse, Toulouse